CLINICAL TRIAL: NCT06063954
Title: A Randomized Trial Comparing Two Electroacupuncture Waveforms for Different Severity Groups of Bell Palsy
Brief Title: Two Electroacupuncture Waveforms for Different Severity Groups of Bell Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Jing Sun, Deputy Chief physician of Traditional Chinese Medicine, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZY-ZJ-KY-23071-01
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Bell Palsy
Keywords: Bell palsy; Acupuncture treatment; Clinical study
MeSH Terms: conditions — Bell Palsy | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-frequency continuous wave group (Experimental): Low-frequency continuous wave EA In each treatment session, the subjects will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 2Hz continuous wave will be used for 20 min.
  Interventions: Other: electroacupuncture
- Intermittent wave group (Experimental): Intermittent wave EA In each treatment session, the subjects will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 40Hz intermittent wave will be used for 20 min.
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — Electroacupuncture (EA) is a form of acupuncture in which a weak electric current is passed through the acupuncture needles into acupoints in the skin.

SUMMARY:
Bell palsy (BP) is the most common cause of acute facial palsy, which leads to functional and esthetic disturbances for patients and results in a lowered quality of life. Electroacupuncture (EA) received attention as an alternative and complementary treatment method. The low-frequency continuous wave EA and the intermittent wave EA have been used in the management of BP. The aim of this study is to compare the efficacy and safety of these two electroacupuncture waveforms for different severity groups of BP.

DETAILED DESCRIPTION:
The investigators will recruit 60 patients with BP whose ENoG test indicate a mild to moderate facial nerve damage, as indicated by the ratio of amplitude of the compound muscle action potential (CMAP) of the affected side comparing to normal side is 20% or higher. And the investigators will recruit 60 patients with BP whose ENoG test indicate a severe damage, as indicated by the ratio of amplitude of the CMAP of the affected side comparing to normal side is less than 20%. Both the two types of patients will be randomly divided into either the low-frequency continuous wave group, or the intermittent wave group, and receive 4 weeks treatment. The primary outcomes is change from baseline score of the Facial Nerve Grading System 2.0. The secondary outcomes are change from baseline score of the Sunnybrook grading scale, and change from baseline value of the amplitude of the CMAP of the affected side in the ENoG test.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as BP by specialist.
2. The score of FNGS 2.0 ≥ 15 at the day 21 since the onset of BP.
3. 18 years ≤ age ≤ 65 years.
4. Received prednisolone within 72 hours since initial symptoms of BP, the prednisolone dose used was 60 mg per day for 5 days and then reduced by 10 mg per day.
5. Signed informed consent and volunteered to participate in this study.

Exclusion Criteria:

1. Facial palsy caused by other diseases or injury.
2. Ramsey-Hunt syndrome.
3. Bilateral facial palsy.
4. History of previous facial palsy.
5. Manifesting facial spasm, facial synkinesis or contracture at day 21 since the onset of BP.
6. History of surgery on face.
7. Combined with uncontrolled diabetes mellitus, uncontrolled hypertension, serious heart, liver, kidney damage or cognitive impairment, aphasia, mental disorders.
8. Installing pacemakers.
9. Pregnant and lactating patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline score of the Facial Nerve Grading System 2.0 | Baseline, the end of week 4
  Evaluation of the facial nerve function using the Facial Nerve Grading System 2.0 (FNGS 2.0). In the FNGS 2.0, the minimal score is 4, which indicates normal function, and the maximal score is 24, which indicates the worst function.

SECONDARY OUTCOMES:
Change from Baseline score of the Sunnybrook grading scale. | Baseline, the end of week 4
  Evaluation of the facial nerve function using the Sunnybrook grading scale. The Sunnybrook grading scale includes 3 subscales, which are the resting symmetry subscale, the symmetry of voluntary movement subscale, and the synkinesis subscale. Change from baseline score of each subscale and change from baseline of the composite score will be calculated.
Change from Baseline value of the amplitude of the compound muscle action potential (CMAP) of the affected side in the ENoG test. | Baseline, the end of week 4
  The compound motor action potential (CMAP) represents the summated action potentials of all stimulated motor endplates and potentially reflects muscle hypertrophy and increased muscle contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sun, MD, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - The Third Affiliated hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Hangzhou First People' s Hospital, Hangzhou, Hangzhou, Zhejing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu ZD, He JB, Guo SS, Yang ZX, Shen J, Li XY, Liang W, Shen WD. Effects of electroacupuncture therapy for Bell's palsy from acute stage: study protocol for a randomized controlled trial. Trials. 2015 Aug 25;16:378. doi: 10.1186/s13063-015-0893-9. PMID 26303741
- [Background] Xu SB, Huang B, Zhang CY, Du P, Yuan Q, Bi GJ, Zhang GB, Xie MJ, Luo X, Huang GY, Wang W. Effectiveness of strengthened stimulation during acupuncture for the treatment of Bell palsy: a randomized controlled trial. CMAJ. 2013 Apr 2;185(6):473-9. doi: 10.1503/cmaj.121108. Epub 2013 Feb 25. PMID 23439629
- [Background] Kim SH, Ryu EW, Yang CW, Yeo SG, Park MS, Byun JY. The prognostic value of electroneurography of Bell's palsy at the orbicularis oculi versus nasolabial fold. Laryngoscope. 2016 Jul;126(7):1644-8. doi: 10.1002/lary.25709. Epub 2015 Oct 15. PMID 26466560
- [Background] Baugh RF, Basura GJ, Ishii LE, Schwartz SR, Drumheller CM, Burkholder R, Deckard NA, Dawson C, Driscoll C, Gillespie MB, Gurgel RK, Halperin J, Khalid AN, Kumar KA, Micco A, Munsell D, Rosenbaum S, Vaughan W. Clinical practice guideline: Bell's palsy. Otolaryngol Head Neck Surg. 2013 Nov;149(3 Suppl):S1-27. doi: 10.1177/0194599813505967. PMID 24189771
- [Background] Marotta N, Demeco A, Inzitari MT, Caruso MG, Ammendolia A. Neuromuscular electrical stimulation and shortwave diathermy in unrecovered Bell palsy: A randomized controlled study. Medicine (Baltimore). 2020 Feb;99(8):e19152. doi: 10.1097/MD.0000000000019152. PMID 32080092
- [Background] Gokce Kutuk S, Ozkan Y, Topuz MF, Kutuk M. The Efficacy of Electro-Acupuncture Added to Standard Therapy in the Management of Bell Palsy. J Craniofac Surg. 2020 Oct;31(7):1967-1970. doi: 10.1097/SCS.0000000000006537. PMID 32472874
- [Background] Vrabec JT, Backous DD, Djalilian HR, Gidley PW, Leonetti JP, Marzo SJ, Morrison D, Ng M, Ramsey MJ, Schaitkin BM, Smouha E, Toh EH, Wax MK, Williamson RA, Smith EO; Facial Nerve Disorders Committee. Facial Nerve Grading System 2.0. Otolaryngol Head Neck Surg. 2009 Apr;140(4):445-50. doi: 10.1016/j.otohns.2008.12.031. PMID 19328328
- [Derived] Bian Z, Wang J, Fang F, Yu B, Shi Y, Wan Y, Hong M, Ji C, Shao X, Liang Y, Fang J, Sun J. Study protocol for a randomized trial comparing two electroacupuncture waveforms for different severity groups of Bell palsy. Front Neurol. 2024 Nov 20;15:1471605. doi: 10.3389/fneur.2024.1471605. eCollection 2024. PMID 39634773